CLINICAL TRIAL: NCT01572610
Title: A Phase 2 GFR Measuring Study of RTA 402 in CKD Patients With Type 2 Diabetes Mellitus
Brief Title: A Glomerular Filtration Rate (GFR) Measuring Study of RTA 402 in Chronic Kidney Disease (CKD) Patients With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTA 402-004
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes
Keywords: CKD patients with type 2 diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RTA 402 (Experimental)
  Interventions: Drug: RTA 402

INTERVENTIONS:
Drug: RTA 402 — once a day, oral administration

SUMMARY:
A Phase 2 glomerular filtration rate (GFR) measuring study of RTA 402 in Chronic kidney disease (CKD) patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
An exploratory study to investigate the effects of RTA 402 on glomerular filtration rate in CKD patients with type 2 diabetes mellitus.

To evaluate the safety of RTA 402.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients with type 2 diabetes mellitus
* Patients whose eGFR levels are eligible for this study
* Patients being treated with stable dose of ACE inhibitors and/or ARB etc.

Exclusion Criteria:

* Patients with Type 1 diabetes
* Patients with known non-diabetic renal disease
* Patients with a history of renal transplantation
* Patients with mean SBP > 160 mmHg or mean DBP > 90 mmHg
* Patients with HbA1C > 10%
* Patients with cardiovascular disease specified in the study protocol
* Patients for whom Inulead® injection is contraindicated etc.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Efficacy: glomerular filtration rate measured by inulin clearance | Up to 16 weeks
  Individual subjects' change from baseline in GFR measured by inulin clearance will be evaluated.
Adverse Event collection and assessment | Up to 16 weeks
  Adverse Event collection

CONTACTS AND LOCATIONS:
Locations (1):
- Koga, Ibaraki, Japan